CLINICAL TRIAL: NCT02041832
Title: Detection of Subclinical Atrial Fibrillation in High Risk Patients (> 65 Years, Hypertension, Diabetes Mellitus) Using Implantable Loop Recorder
Brief Title: Detection of Subclinical Atrial Fibrillation in High Risk Patients Using Implantable Loop Recorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axel Brandes (Other)
Responsible Party: Sponsor-Investigator, Axel Brandes, Associate Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ILR-Afib-study; S-20130062 (Other: Videnskabsetisk Komité for Region Syddanmark)
Record Dates: First submitted 2013-11-28; First posted 2014-01-22 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Arterial Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Holter monitoring (Other): Screening of patients with older age, arterial hypertension and diabetes for paroxysmal atrial fibrillation by using conventional Holter monitoring
  Interventions: Other: Conventional Holter monitoring
- Implantable loop recorder (Other): Screening of patients with older age, arterial hypertension and diabetes mellitus for paroxysmal atrial fibrillation by using an implantable loop recorder
  Interventions: Device: Implantable loop recorder

INTERVENTIONS:
Other: Conventional Holter monitoring — Patients undergo 72h Holter monitoring
  Arms: Holter monitoring
Device: Implantable loop recorder — Implantation of loop recorder with follow-up by remote monitoring
  Other Names: REVEAL XT
  Arms: Implantable loop recorder

SUMMARY:
Using implantable loop recorder the investigators wish to detect atrial fibrillation in high risk patients and compare it to the results using conventional Holter monitoring. The hypothesis is that 10-15% of high risk patients have subclinical atrial fibrillation. The investigators want to detect those people so they can receive appropriate anticoagulation treatment. The patients will get a comprehensive workup including ecg, echocardiography and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* age > 65 years
* arterial hypertension (at least dual treatment)
* diabetes mellitus (oral antidiabetics or insulin)

Exclusion Criteria:

* known atrial fibrillation
* ischaemic heart disease
* Current anticoagulation treatment
* Ejection fraction <45 %
* significant valvular heart disease
* previous stroke/transient ischemic attack
* peripheral arterial disease
* end stage renal disease
* thyreotoxicosis

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
First episode of atrial fibrillation | 1 year

SECONDARY OUTCOMES:
Correlation between echocardiographic parameters and incidence of atrial fibrillation | 1 year

OTHER OUTCOMES:
Correlation between biomarkers and incidence of atrial fibrillation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Axel Brandes, Assoc. Prof., Study Director — Odense University Hospital/University of Southern Denmark
Locations (1):
- Haderslev Hospital, Haderslev, Denmark

REFERENCES:
- [Derived] Philippsen TJ, Christensen LS, Hansen MG, Dahl JS, Brandes A. Detection of Subclinical Atrial Fibrillation in High-Risk Patients Using an Insertable Cardiac Monitor. JACC Clin Electrophysiol. 2017 Dec 26;3(13):1557-1564. doi: 10.1016/j.jacep.2017.06.020. Epub 2017 Nov 6. PMID 29759838